CLINICAL TRIAL: NCT04725123
Title: Bezlotoxumab Yielded Outcomes by Addressing Personalized Needs in Clostridioides Difficile Infection: Study Phase 1
Brief Title: Addressing Personalized Needs in Clostridioides Difficile Infection
Acronym: BEYOND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hellenic Institute for the Study of Sepsis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BEYOND1
Record Dates: First submitted 2021-01-25; First posted 2021-01-26 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Clostridioides Difficile Infection
Keywords: Clostridioides difficile; Microbiome; Prediction; Unfavorable outcome
MeSH Terms: conditions — Clostridium Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Clostridioides difficile infection (Experimental): Stool of patients with Clostridioides difficile infection that will be subject to microbiome analysis. Comparisons will be done between patients with favorable and unfavorable outcome
  Interventions: Diagnostic Test: Microbiome analysis

INTERVENTIONS:
Diagnostic Test: Microbiome analysis — Stool microbiome analysis of 16S rRNA sequencing to an anticipated number of 8,000,000 reads

SUMMARY:
BEYOND is aiming to demonstrate how by enrichment of the available SPECIFY score, patients at great likelihood for CDI with unfavorable outcome are early detected

DETAILED DESCRIPTION:
In a previous project, following GWAS analysis of the DNA and measurement of serum biomarkers coming from 134 patients a prediction score named SPECIFY was developed. The SPECIFY score comprises four elements: low hemoglobin, increased urea, increased IL-8 and carriage of G alleles of rs2091172. The score has 80% positive predictive value and 95.8% specificity for the early detection of unfavorable outcome but the sensitivity is low. Unfavorable outcome is defined as any of: presentation or progression into severe CDI, relapse; and death. Stool samples of day 1 before start of therapy of the patients are stored refrigerated. Microbiome analysis will be done aiming to the integration of the Shannon diversity index to the already developed score in order to improve sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Age more than or equal to 18 years
* Both genders
* Diarrhea defined as at least 3 episodes of unformed stools in the last 24hours according to the Bristol stool chart
* Presence of C.difficile in stool. This is defined as any stool sample positive for the presence of glutamate dehydrogenase (GDH) and for the presence of toxin A and/or B.

Exclusion Criteria:

• No exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2021-01-26 (Actual); Primary Completion 2022-03-27 (Actual); Study Completion 2022-03-27 (Actual)

PRIMARY OUTCOMES:
Prediction of unfavorable outcome | 40 days
  Sensitivity of the BEYOND score to predict unfavorable outcome of patients with infection by Clostridioides difficile

SECONDARY OUTCOMES:
Diagnostic PCR reaction in stool | 40 days
  Development of one RT-PCR reaction informing of the predominance of bacterial generum causing low microbiome diversity associated with the unfavorable outcome of CDI.

CONTACTS AND LOCATIONS:
Overall Officials: Evangelos J Giamarellos-Bourboulis, MD, PhD, Study Chair — National and Kapodistrian University of Athens
Locations (1):
- 4th Department of Internal Medicine, ATTIKON University General Hospital, Athens, Greece

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared with other investigators after the end of the study.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: After the end of the study
Access Criteria: Signed contract for data sharing with the study Sponsot

REFERENCES:
- [Derived] Psarrakis C, Tziolos NR, Matzarakis V, Kumar V, Stylianakis E, Sidiropoulou C, Tasouli E, Iliopoulou K, Samarkos M, Metallidis S, Georgiadou S, Akinosoglou K, Bolanou A, Hatziagelaki E, Kostaki A, Panagopoulos P, Toutouzas K, Milionis H, Adamis G, Poulakou G, Lada M, Skoutelis A, Alexiou Z, Symbardi S, Chrysos G, Netea MG, Giamarellos-Bourboulis EJ. A randomized controlled trial of precision bezlotoxumab treatment for Clostridioides difficile infection. Cell Rep Med. 2026 Jan 20;7(1):102533. doi: 10.1016/j.xcrm.2025.102533. Epub 2026 Jan 2. PMID 41483804